CLINICAL TRIAL: NCT01803893
Title: Preimplantation Factor (PIF): Prognostic Value of a Non-invasive Embryo Viability Biomarker Detection in Culture Media Followed by Single Embryo Transfer - Correlation With Live Birth.
Brief Title: Prognostic Value of PIF Detection in Embryo Culture Media Correlation With Pregnancy Outcome
Acronym: PIF-SET1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: BioIncept LLC (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: BioIncept LLC-1; GFI Merck Serono 2012 (Other Grant/Funding Number: GFI-1)
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Pregnancy; Fertility
Keywords: In vitro fertilization; implantation; miscarriage; live birth
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — embryo culture media
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Embryo culture media: measurement using immunoassay
- maternal serum: measurement by immunoassay

SUMMARY:
PIF: biomarker of successful implantation To overcome the poor reproductive potential of embryos generated during in vitro fertilization cycles and the lack of markers enabling the identification of the most competent ones, it is common to transfer multiple embryos. However this practice is associated with the risks of multi-fetal pregnancies and high morbidity/mortality. Ideally, the availability of a marker specifically produced by viable embryos would permit the transfer of a single embryo (SET) without affecting the chances of pregnancy and, most importantly, capable to drastically reduce multiple pregnancies after IVF. In preliminary work, we demonstrated that no pregnancy resulted following the transfer of embryos where PIF was undetectable in culture media.(Keramitsoglou, T et al. ASRI Meeting, Hamburg, 2012) Using a non-invasive method of detection of PIF in the media surrounding the embryo will be correlated to live birth following single embryo transfer. By selecting only viable embryos, it will reduce the need for multiple IVF cycles, increase the rate of pregnancy outcome associated with SET, and will minimize multi-fetal pregnancy that has very high medical and societal costs both in pregnancy and after delivery.

DETAILED DESCRIPTION:
The aim of the proposed project is to investigate a non invasive biomarker, PIF (PreImplantation Factor), a 15amino acid peptide (MVRIKPGSANKPSDD) secreted only by viable embryos and placenta (Stamakin et al. RBE 2011).

PIF positive embryos will be able to grow to blastocyst stage and PIF levels could be a marker of progressive pregnancy. We will measure PIF levels in IVF culture media before embryo transfer to correlate IVF pregnancy with PIF levels. Our objective will be to define PIF as a biomarker for viable embryos in order to increase IVF success rates following SET. PIF levels will be retrospectively evaluated after 500 SET.

Our four reproductive centres perform about 200 SET per year and more than 500 in vitro fertilizations.

For women selected for a SET, PIF levels will be evaluated in all embryo culture media, and later at one and two weeks after each transfer of fresh or thawed frozen embryos in maternal serum. Embryo transfers will be done blinded to PIF results. SET or MET will be based on clinical evaluation and conventional embryo criteria. For these women, PIF will be also evaluated and compared with βhCG level on maternal serum.

PIF assessment will be performed using specific antibody marked with a fluorescent dye, in Luminex reader.

Specific Aim One will allow us to evaluate:

* PIF predictive value on implantation rate
* PIF predictive value on pregnancy Methodology All women will be fully informed and a written consent to participate in the study will be duly obtained.

In vitro procedure Oocytes were retrieved after natural cycle or after ovarian hyperstimulation which will be performed using the modified long protocol. Collected oocytes will be fertilized by classic IVF or ICSI. Fertilization will be confirmed by the observation of 2 pronuclei and two polar bodies, after 16-18 hours. Fertilized oocytes will be cultured in 60μl of culture media under oil. Embryo transfer will be performed 72 hours after IVF or ICSI procedure (at day D3) without PIF result. Before transfer, embryo quality will be scored according to number of cells, kinetic of cleavage and fragmentation rate. For women who will have a SET, according to clinical criteria (Age, FSH level, etc…) remaining good quality embryos will be frozen and thawed after uterine preparation in further attempts. All remaining culture supernatants (50-60μl) will be collected, transferred to 8-strip 0.2ml tubes and stored to -80C until they will test for PIF (M) Maternal serum retrieval

Maternal serum will be collected:

* before oocytes retrieval in course of a serum control of ovarian hyperstimulation (S0)
* one week after transfer (S1)
* two week after transfer during serial human β-chorionic gonadotrophin measurements (S2) PIF level evaluation PIF levels in culture supernatants and in maternal serum will be measured retrospectively, using a bead-based competitive assay for use in the Luminex 200 IS system. Results presented as median fluorescence intensity (MFI). PIF levels were derived from standard curve using a 5-parameter logistics curve. The threshold of detection was established by measuring the background from culture media or maternal serum alone, using mean+2SD as a cut off (18.7ng/ml).

Analysis Correlate PIF detection in embryo serum with embryo viability. Results of PIF detection in embryo supernatants will be correlated with pregnancy outcome.

Comparison with embryo selection by PIF+ vs PIF- embryos, using morphology alone, and by morphology combined with PIF presence.

Comparisons between groups will be performed using chi-square analysis and p<0.05 will be considered as statistically significant.

Inclusion/exclusion criteria

Inclusion criteria:

All women included in our centers for classical IVF or ICSI, who will sign the written consent to participate in the study. PIF level evaluation in culture media (M) and pregnancy prognosis (S1 and S2) will be done only for women with SET.

Exclusion criteria Women who will refuse to participate in the program. Planned assessments (time and events table) The overall project is planned to be carried out through five steps work plan in which we will investigate the use of PIF as a biomarker for better embryo selection (only women with SET will be included) and as a early pregnancy marker in maternal serum.

ELIGIBILITY:
Inclusion criteria:

All women included in our centers for classical IVF or ICSI, who will sign the written consent to participate in the study. PIF level evaluation in culture media (M) and pregnancy prognosis (S1 and S2) will be done only for women with SET.

Exclusion criteria Women who will refuse to participate in the program.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Infertile women attending IVF center who undergo in vitro fertilization in order to achieve pregnancy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Detection of PIF in early pregnancy maternal serum | end of pregnancy
  Following PIF positive single embryo transfer, patients' pregnancy will be monitored by standard methods. This includes: blood tests and ultrasound until pregnancy viability has been established. The number of patients that fail to implant or end up in implantation failure (ie chemical pregnancy), miscarriage, gestational sac will be recorded.

SECONDARY OUTCOMES:
Correlation between PIF positive and negative embryos and early pregnancy events | end of pregnancy
  SET embryo transfers will be performed blinded, unrelated to PIF results. Subsequent to SET, the embryo culture media will be tested for presence/absence of PIF and documented. Following transfer, patients' pregnancy will be monitored by standard methods. This includes: blood tests and ultrasound to determine embryo viability.
Correlation between PIF positive and negative embryos and late pregnancy events | end of pregnancy
  SET embryo transfers will be performed blinded, unrelated to PIF results. Subsequent to SET, the embryo culture media will be tested for presence/absence of PIF and documented. Following transfer, patients' pregnancy will be monitored by standard methods. Once viability is established by standard methods, patients will be followed throughout pregnancy until eventual delivery. Premature delivery, high risk pregnancy events will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Eytan R Barnea, MD, FACOG, Study Chair — BioIncept LLC
Locations (5):
- Yale Women and Children's Center for Blood Disorders & Yale Fertility Center, New Haven, Connecticut, United States
- France (3):
  - Poissy St Germain Hospital, Poissy, Cedex
  - Lab Clement - Seine St. Denis Hospital, Le Blanc Mesnil, Paris
  - Versailles St. Quentin University, Poissy
- Helena Venizelou Hospital, Athens, Greece